CLINICAL TRIAL: NCT00368992
Title: A Phase II Trial of Combination Carboplatin, Paclitaxel, Cetuximab and Bevacizumab (NSC-704865) Followed By Cetuximab and Bevacizumab in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: S0536: Cetuximab, Paclitaxel, Carboplatin, and Bevacizumab in Treating Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02903; S0536; U10CA032102 (NIH)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2013-02

CONDITIONS: Adenocarcinoma of the Lung; Adenosquamous Cell Lung Cancer; Bronchoalveolar Cell Lung Cancer; Large Cell Lung Cancer; Recurrent Non-small Cell Lung Cancer; Squamous Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Paclitaxel; Taxes; Bevacizumab

ARMS (1):
- Treatment (cetuximab, paclitaxel, bevacizumab) (Experimental): INDUCTION THERAPY: Patients receive cetuximab IV over 1-2 hours on days 1, 8, and 15 and paclitaxel IV over 3 hours, carboplatin IV over 30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive cetuximab IV over 1 hour on days 1, 8, and 15 and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cetuximab; Drug: paclitaxel; Biological: bevacizumab

INTERVENTIONS:
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF

SUMMARY:
Monoclonal antibodies, such as cetuximab and bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Bevacizumab may stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving cetuximab together with paclitaxel, carboplatin, and bevacizumab may kill more tumor cells. This phase II trial is studying how well giving cetuximab together with paclitaxel, carboplatin, and bevacizumab works in treating patients with advanced non-small cell lung cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the frequency and severity of hemorrhage toxicities in patients with advanced non-small cell lung cancer treated with the combination of carboplatin, paclitaxel, cetuximab and bevacizumab followed by therapy with cetuximab and bevacizumab.

SECONDARY OBJECTIVES:

I. To evaluate progression-free and overall survival, response rate (confirmed plus unconfirmed, complete plus partial), and frequency and severity of non-hemorrhage toxicities in this group of patients treated with this regimen.

II. To perform molecular correlative studies on patient tissue to investigate in an exploratory manner potential predictors of efficacy.

OUTLINE: This is a multicenter study.

INDUCTION THERAPY: Patients receive cetuximab IV over 1-2 hours on days 1, 8, and 15 and paclitaxel IV over 3 hours, carboplatin IV over 30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive cetuximab IV over 1 hour on days 1, 8, and 15 and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically proven newly diagnosed selected stage IIIB (T4 lesion due to malignant pleural effusion) or stage IV, advanced primary non-small cell lung cancer (adenocarcinoma, large cell carcinoma, or unspecified) or recurrent disease after previous surgery and/or irradiation; patients with tumors having squamous cell components > 50% are not eligible
* Patients with known brain metastases are not eligible; all patients must have a pretreatment CT or MRI scan of the brain to evaluate for CNS disease within 42 days prior to registration
* Patients may have measurable or non-measurable disease documented by CT, MRI, X-ray or physical exam; measurable disease must be assessed within 28 days prior to registration; pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease; non-measurable disease must be assessed within 42 days prior to registration; all disease must be assessed and documented on the Baseline Tumor Assessment Form (Form #848)
* Patients must not have received any prior systemic chemotherapy or biologic therapy for non-small cell lung cancer; patients must not have received any adjuvant therapy for non-small cell lung cancer
* Prior radiation is permitted; however, at least three weeks must have elapsed since the completion of prior radiation therapy and patients must have recovered from all associated toxicities at time of registration; measurable or non-measurable disease must be outside the previous radiation field or a new lesion must be present
* At least four weeks must have elapsed since surgery (thoracic or other major surgeries) and patients must have recovered from all associated toxicities at the time of registration; measurable disease must be present outside the area of surgical resection; there must be no anticipation of need for major surgical procedures during protocol treatment
* Patients must not have received prior cetuximab, ZD1839, erlotinib or other investigational agents that target the EGFR pathway; patients must not have received prior VEGF-related agents; patients must not have received prior chimerized or murine monoclonal antibody therapy or have documented presence of human anti-mouse antibodies (HAMA)
* ANC >= 1,500/mcl
* Platelet count >= 100,000/mcl
* Hemoglobin >= 9 mg/dl
* Patients must have a serum creatinine =< institutional upper limit of normal (IULN) AND calculated or measured creatinine clearance >= 50 cc/min using the Cockroft-Gault Formula
* Urine protein must be screened by urine analysis for Urine Protein Creatinine (UPC) ratio; for UPC ratio > 0.5, 24-hour urine protein must be obtained and the level must be < 1,000 mg for patient enrollment
* Serum bilirubin =< 2 x IULN
* Either SGOT or SGPT =< 2 x IULN (if both SGOT and SGPT are done, both must be =< 2 x IULN)
* International Normalized Ratio (INR) =< 1.5; patients must not be taking full-dose anticoagulation therapy; patients may be enrolled initially if they are on low-dose warfarin (i.e., 1 mg daily)
* All patients must have a Zubrod performance status of 0 - 1
* Correlative science studies: institutions must have received IRB approval of S9925 (the Lung Cancer Specimen Repository); patients must be offered participation in S9925; with the patient's consent, blood, plasma and tissue will be submitted for testing via S9925; patients must be registered separately to S9925 in order for institutions to receive credit for specimen submissions
* Patients must not have had hemoptysis >= 1/2 teaspoon within 3 months prior to registration
* Patients must not have >= grade 2 symptomatic neuropathy-sensory (National Cancer Institute [NCI] Common Terminology Criteria Version 3.0)
* Patients must not have documented evidence of acute hepatitis or have an active or uncontrolled infection
* Patients must not have the following: history (within past 6 months) of CVA, myocardial infarction or unstable angina; uncontrolled hypertension; New York Heart Association grade 2 or greater congestive heart failure; serious cardiac arrhythmia requiring medication; or clinically significant peripheral vascular disease
* Patients must not have had an open biopsy or significant traumatic injury within 28 days prior to registration; patients must not have had a core biopsy within 7 days prior to registration
* Patients must not have serious or non-healing wound, ulcer or bone fracture
* Patients must not have history of abdominal fistula, gastrointestinal perforation or intraabdominal abscess within 28 days prior to registration
* Patients must have no known hypersensitivity of Chinese hamster ovary cell products or other recombinant human antibodies
* Patients must not have evidence of bleeding diathesis or coagulopathy
* Patients must be willing to provide prior smoking history as required on the S0536 Prestudy Form (Form #54655)
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* Pregnant or nursing women are not eligible for this trial; women/men of reproductive potential must not participate unless they have agreed to use an effective contraceptive method during protocol treatment and for at least 6 months following completion of bevacizumab treatment
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and ID number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Kim, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Carboplatin, Paclitaxel, Cetuximab, and Bevacizumab: This was a single arm Phase II trial. Patients were treated with induction therapy cetuximab IV over 1-2 hours on days 1, 8, and 15 and paclitaxel IV over 3 hours, carboplatin IV over 30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Patients who were not removed due to unacceptable toxicity or disease progression were then treated with maintenance therapy cetuximab IV over 1 hour on days 1, 8, and 15 and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Carboplatin, Paclitaxel, Cetuximab, and Bevacizumab
Started | 110
Completed | 0
Not Completed | 110
Not completed — Ineligible | 5
Not completed — Refused treatment | 3
Not completed — Lack of Efficacy | 63
Not completed — Adverse Event | 26
Not completed — Death | 4
Not completed — Other | 9

BASELINE CHARACTERISTICS:
Groups:
- Carboplatin, Paclitaxel, Cetuximab, and Bevacizumab: This was a single arm Phase II trial. Patients were treated until progression.
Arm/Group | Carboplatin, Paclitaxel, Cetuximab, and Bevacizumab
Number analyzed (Participants) | 102
Age, Continuous [Median (Full Range); unit: years] | 64 [42 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 52

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With Grade 4 (i.e. Life-threatening) Hemorrhage Toxicities Related to Protocol Treatment.
Description: All patients who received protocol treatment were assessed for adverse events per the NCI Common Terminology Criteria for Adverse Events, Version 3.0. We counted the number of patients who reported at least one Grade 4 (i.e. life-threatening) hemorrhage adverse event that was possibly, probably, or definitely related to the study treatment.
Time Frame: Every week until removed from protocol therapy, up to 3 years.
Population: Eligible patients who received protocol treatment were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carboplatin, Paclitaxel, Cetuximab, and Bevacizumab
Number analyzed (Participants) | 102
percentage of participants | 2 [0 to 7]

2. Secondary Outcome: Progression-Free Survival
Description: From data of registration to date of disease progression (as defined by RECIST, i.e. a 20% increase in the sum of the longest diameters of target lesions, or unequivocal progression ina non-target lesion in the opinion of the treating investigator, or the appearance of new lesions), symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression-free were censored at the date of last contact.
Time Frame: Every 6 weeks until disease progression. After 9 months, every 12 weeks until disease progression, up to 3 years.
Population: Eligible patients who received protocol treatment were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin, Paclitaxel, Cetuximab, and Bevacizumab
Number analyzed (Participants) | 102
Months | 7 [6 to 8]

3. Secondary Outcome: Overall Survival
Description: From date of enrollment to date of death due to any cause. Patients last known to be alive were censored at date of last contact.
Time Frame: Once a week, up to 3 years.
Population: Eligible patients who received protocol treatment were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin, Paclitaxel, Cetuximab, and Bevacizumab
Number analyzed (Participants) | 102
months | 15 [11 to 21]

4. Secondary Outcome: Response Rate
Description: Confirmed and unconfirmed complete and partial responses per RECIST in the subset of patients with at least one target lesion assessed by CT or MRI. A complete response (CR) was defined as disappearance of all disease, including non-target lesions. A partial response (PR) was defined as a >= 30% decrease in the sum of the longest diameters of all target lesions. A CR or PR was confirmed if documented a second time at least 4 weeks after the first documentation.
Time Frame: Every 6 weeks while on protocol treatment, up to 3 years.
Population: Eligible patients who received protocol treatment and who had measurable disease (as defined by RECIST) at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carboplatin, Paclitaxel, Cetuximab, and Bevacizumab
Number analyzed (Participants) | 95
percentage of participants | 56 [44 to 65]

ADVERSE EVENTS:
Time Frame: Weekly while on protocol treatment.
Arm/Group | Carboplatin, Paclitaxel, Cetuximab, and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 51/102
Other Adverse Events (participants affected / at risk) | 101/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin, Paclitaxel, Cetuximab, and Bevacizumab (N=102)
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Hemoglobin (Blood and lymphatic system disorders) | 1
Cardiac-ischemia/infarction (Cardiac disorders) | 1
Left ventricular diastolic dysfunction (Cardiac disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Ventricular arrhythmia - Ventricular tachycardia (Cardiac disorders) | 1
Ocular/Visual-Other (Specify) (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 5
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Death not associated with CTCAE term - Death NOS (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6
Sudden death (General disorders) | 1
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 1
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 1
Inf (clin/microbio) w/Gr 3-4 neuts - Colon (Infections and infestations) | 1
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 4
Inf (clin/microbio) w/Gr 3-4 neuts - Sinus (Infections and infestations) | 1
Inf (clin/microbio) w/Gr 3-4 neuts - UTI (Infections and infestations) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Joint (Infections and infestations) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 3
Inf w/normal ANC or Gr 1-2 neutrophils - Mid ear (Infections and infestations) | 1
Infection with unknown ANC - Blood (Infections and infestations) | 1
Leukocytes (total WBC) (Investigations) | 3
Lymphopenia (Investigations) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 16
Platelets (Investigations) | 2
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 7
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal/Soft Tissue-Other (Specify) (Musculoskeletal and connective tissue disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 2
Pain - Buttock (Musculoskeletal and connective tissue disorders) | 1
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 2
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
CNS cerebrovascular ischemia (Nervous system disorders) | 1
Neuropathy: motor (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 1
Ocular/Visual-Other (Specify) (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Syncope (fainting) (Nervous system disorders) | 2
Vaginitis (not due to infection) (Reproductive system and breast disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 9
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pain - Pleura (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Phlebitis (including superficial thrombosis) (Vascular disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin, Paclitaxel, Cetuximab, and Bevacizumab (N=102)
Hemoglobin (Blood and lymphatic system disorders) | 58
Vision-blurred vision (Eye disorders) | 6
Constipation (Gastrointestinal disorders) | 57
Diarrhea (Gastrointestinal disorders) | 45
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 7
Heartburn/dyspepsia (Gastrointestinal disorders) | 15
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 36
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 21
Nausea (Gastrointestinal disorders) | 53
Pain - Abdomen NOS (Gastrointestinal disorders) | 11
Pain - Oral cavity (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 25
Edema: limb (General disorders) | 10
Fatigue (asthenia, lethargy, malaise) (General disorders) | 88
Pain - Chest/thorax NOS (General disorders) | 10
Pain-Other (Specify) (General disorders) | 14
Rigors/chills (General disorders) | 6
Allergic reaction/hypersensitivity (Immune system disorders) | 14
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 11
Infection-Other (Specify) (Infections and infestations) | 8
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 22
AST, SGOT (Investigations) | 22
Alkaline phosphatase (Investigations) | 31
Bilirubin (hyperbilirubinemia) (Investigations) | 8
Creatinine (Investigations) | 6
Leukocytes (total WBC) (Investigations) | 52
Lymphopenia (Investigations) | 9
Metabolic/Laboratory-Other (Specify) (Investigations) | 6
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 62
Platelets (Investigations) | 40
Weight loss (Investigations) | 40
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 30
Anorexia (Metabolism and nutrition disorders) | 43
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 31
Dehydration (Metabolism and nutrition disorders) | 17
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 56
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 11
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 50
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 11
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 21
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 29
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 8
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 14
Pain - Back (Musculoskeletal and connective tissue disorders) | 19
Pain - Bone (Musculoskeletal and connective tissue disorders) | 17
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 9
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 20
Pain - Joint (Musculoskeletal and connective tissue disorders) | 32
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 24
Dizziness (Nervous system disorders) | 21
Neuropathy: motor (Nervous system disorders) | 11
Neuropathy: sensory (Nervous system disorders) | 76
Pain - Head/headache (Nervous system disorders) | 13
Taste alteration (dysgeusia) (Nervous system disorders) | 25
Insomnia (Psychiatric disorders) | 19
Mood alteration - anxiety (Psychiatric disorders) | 15
Mood alteration - depression (Psychiatric disorders) | 19
Proteinuria (Renal and urinary disorders) | 13
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 27
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 44
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 27
Mucositis/stomatitis (functional/symp) - Pharynx (Respiratory, thoracic and mediastinal disorders) | 7
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 8
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 21
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 16
Dry skin (Skin and subcutaneous tissue disorders) | 26
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 50
Nail changes (Skin and subcutaneous tissue disorders) | 6
Pruritus/itching (Skin and subcutaneous tissue disorders) | 22
Rash/desquamation (Skin and subcutaneous tissue disorders) | 31
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 78
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 9
Hypertension (Vascular disorders) | 25
Hypotension (Vascular disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less